CLINICAL TRIAL: NCT06982703
Title: Evaluation of Butyrate, Zinc and Vitamine D Effect on Microbiota Modulation and Prevention of Antibiotic-associated Diarrhea
Brief Title: Evaluation of Butyrate Effect on Diarrhea
Acronym: DBZ
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5907/AO/24
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: antibiotics, microbiota, diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Vitamin D; Zinc

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, randomized trial, in which the enrolled subjects will be included in one year. After enrolment and written informed consent collection, 50 subjects will be randomized in a 1:1 ratio to Group 1 or Group 2 . During the study supplement administration subjects will be requested to avoid probiotics, while only fermented foods normally consumed will be allowed
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dibuzin (Active Comparator): Group1: 2 capsules/day of DBZ (1 /morning and 1 /evening, away from meals) for 14 gg
  Interventions: Dietary Supplement: Food Supplement DBZ (acronym for: DIBUZIN) containing calcium butyrate, vitamin D and zinc,
- Placebo (Placebo Comparator): Group2: 2 capsules/day of Placebo (1 /morning and 1 /evening, away from meals) for 14 gg
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food Supplement DBZ (acronym for: DIBUZIN) containing calcium butyrate, vitamin D and zinc, — In this prospective pilot study, we plan to evaluate the effects of a Food Supplement DBZ (acronym for: DIBUZIN) containing calcium butyrate, vitamin D and zinc, on the variation of intestinal microbiota and prevention of antibiotic-induced diarrhea, in individuals who have been prescribed antibiotic therapy.
  Arms: Dibuzin
Dietary Supplement: Placebo — The intervention with Placebo involves the intake of a product free of bityrate, zinc and vitD
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effects of a Food Supplement containing calcium butyrate, vitamin D, and zinc, on the variation of intestinal microbiota and prevention of antibiotic-induced diarrhea, in individuals who have been prescribed antibiotic therapy. The main questions it aims to answer is:

Does Dibuzin improve the microbiota composition in patients undergoing antibiotic treatment? Does Dibuzin prevent antibiotic-induced diarrhea? Participants will: - take 2 capsules/day of DBZ (1 /morning and 1 /evening, away from meals) for 14 gg. -Visit the clinic two times ( T0 and at the end), collect three fecal samples, and fill out two questionnaires 3 times.

DETAILED DESCRIPTION:
Antibiotic-associated diarrhea (AAD) is an important morbidity resulting from antibiotic use. AAD is more than a bothersome adverse event of antibiotic treatment; it is associated with prescription noncompliance and overuse of second-line antibiotics. Any antibiotic could potentially cause AAD, but broad-spectrum antibiotics that predominantly target anaerobes and are poorly absorbed, have a higher AAD incidence. Alterations in the diversity of the gut microbiota are believed to underlie the development of antibiotic-associated diarrhea, likewise, micronutrient deficiencies can exacerbate both barrier leak and morbidity.

The use of SCFAs, such as butyrate, along with vitamin D and zinc, each possessing unique properties that contribute to enhancing the microbiota, controlling inflammation, and promoting a healthy intestinal barrier, may be beneficial in the prevention of AAD.

The proposed dietary supplement contains butyrate, vitamin D, and zinc, and is presented as a potential product useful in the prevention of AAD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing antibiotic therapy
* Subjects capable of conforming to the study protocol
* Subjects who have given their free and informed consent

Exclusion Criteria:

* Subjects with untreated food intolerance, i.e. remaining symptomatic despite the withdrawal of the suspected food
* Subjects who become unable to conform to protocol
* Subjects who are continuously taking contact laxatives Subjects who are treated with pre/probiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the variation of gut microbiota composition (microbiota test) | 9 months
  Collection of faecal sample for the assessment of the faecal microbiota composition ( rRNA16S) The 16S rRNA gene is a bacterial ribosomal gene and a part of the 30S subunit which is used in the identification, characterization, and classification of various bacteria. Samples were normalized, pooled, and run on Illumina MiSeq , in order to evaluate the composition of gut microbiota in terms of bacterial diversity ( alfa and beta) and abundance and any variability associated with the treatment.

SECONDARY OUTCOMES:
Evaluation of gastrointestinal symptoms ( VAS scale) | 9 months
  The patient will report the gastrointestinal symptoms on a form ( VAS scale), daily
Assessment of prevention of Antibiotic-associated diarrhea | 9 months
  The patient will report on a form the diarrheal episodes, using a scale from 1 to 10, daily.
Evaluation of psychological state and quality of life ( SF-12) | 9 months
  The patient will report a questionnaire (SF-12) on the quality of life at the visits.

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo V. Savarino, medical doctor, PhD, Principal Investigator — UniPD-AOUP
Locations (1):
- Edoardo V. Savarino, Padua, Italy